CLINICAL TRIAL: NCT03134066
Title: Neurocognitive Features of Patients With Treatment-Resistant Depression
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Staff Psychiatrist, Massachusetts General Hospital
Other Study IDs: 2016P001654
Record Dates: First submitted 2017-04-18; First posted 2017-04-28 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Treatment-resistant depression patients: Subjects with TRD who have been deemed appropriate for (and have decided to receive) clinical, non-research ketamine treatment at the ketamine clinic at Massachusetts General Hospital. As this is an assessment-only observational study, no treatment assignment or randomization procedures will be used.

SUMMARY:
There is an urgent need for novel and effective interventions for treatment-resistant depression (TRD). In previous studies, ketamine has been shown to rapidly reduce depressive symptoms; however, the exact mechanisms of action of ketamine remain unknown. There are some preliminary findings to suggest that ketamine may exert its antidepressant effects through promotion of neurogenesis in the dentate gyrus. The aim of this study is to help delineate the neurocognitive effects of ketamine exposure using a behavioral task (specifically, a pattern separation task) and a battery of other well-established cognitive measures.

This is an assessment-only study, as we will be recruiting subjects to complete an assessment battery at two time points, before and after receiving ongoing ketamine administrations for at least four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. be 18-80 years old
2. be able to read, understand, and provide written informed consent in English,
3. meet criteria for a current moderate/severe (> 14 on QIDS-SR) depressive episode (unipolar or bipolar mood disorder),
4. have a history of > 3 failed antidepressant trials, and be
5. be seeking ketamine ongoing treatment through the ketamine clinic at Massachusetts General Hospital and be deemed appropriate for the clinic.

Exclusion Criteria:

1. Subjects who will not provide consent to neuropsychological testing
2. Subjects who are not deemed appropriate for the ketamine clinic will not be enrolled

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligibility for participants includes those ages 18-80 years old who meet criteria for a moderate/severe (as indicated by a score of > 14 on the QIDS-SR) depressive episode (unipolar or bipolar mood disorder), have a history of at least three failed antidepressant trails, and are seeking non-research ketamine treatment through the ketamine clinic at Massachusetts General Hospital (and are deemed appropriate for treatment at the clinic. Participants must also be able to read, understand, and provide written informed consent in English.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2018-01-17 (Actual)

PRIMARY OUTCOMES:
Change in pattern separation task results | Baseline - post at least 2 weeks on a stable dose of intranasal ketamine
  The pattern separation task is a computer-based behavioral task that captures characteristic of pattern separation processes. Pattern separation is thought to be involved in the process of you finding your car everyday despite being in a different space; this may be dysfunctional in people with depression. The task itself is not an intervention; it is a rapid assessment of putative changes in pattern separation.